CLINICAL TRIAL: NCT03767361
Title: Study the Effect of Blood Transfusion on Oxidant-antioxidant Status in Term and Near-term Neonates
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rania Ali El-Farrash (Other)
Responsible Party: Sponsor-Investigator, Rania Ali El-Farrash, Clinical Professor, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: MS2015
Record Dates: First submitted 2017-08-07; First posted 2018-12-06 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Blood Transfusion Complication; Oxidative Stress
MeSH Terms: conditions — Transfusion Reaction

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fresh PRBCs (Active Comparator): Neonates will receive fresh packed red blood cells transfusion within 7 days of donation
  Interventions: Biological: packed red blood cells transfusion
- Old PRBCs (Active Comparator): Neonates will receive fresh packed red blood cells transfusion older than 7 days yet within the standard range accepted universally will be transfused to this group.
  Interventions: Biological: packed red blood cells transfusion

INTERVENTIONS:
Biological: packed red blood cells transfusion — packed red blood cells transfusion

SUMMARY:
Primary aim is to evaluate the effect of blood transfusion on oxidant-antioxidant status in premature neonates. Secondary aim is to assess the effect of the age of transfused red blood cells on the biological markers of oxidative stress.

DETAILED DESCRIPTION:
Oxidant-antioxidant status will be assessed by measuring total antioxidant capacity (TAC) and malondialdehyde (MDA), as well as antioxidant minerals, in 65 term and near-term neonates.

ELIGIBILITY:
Inclusion Criteria:

* Premature neonates ≤36 weeks in need for blood transfusion.

Exclusion Criteria:

* Critically ill neonates.(perinatal asphaxia,on high setting mechanical ventilation,different types of shock eg ;septic shock and major congenital anomalies)
* Extremely low birth weight neonates(<1000gm birth weight )
* Recipient of blood transfusion before enrollment in the study.
* Neonates planned for exchange transfusion .

Ages: 35 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
malondialdehyde | 2-3 hours posttransfusion
  MDA
total antioxidant capacity | 2-3 hours posttransfusion
  TAC
serum Copper | 2-3 hours posttransfusion
  s.Cu
serum Zinc | 2-3 hours posttransfusion
  s.Zn
serum magnesium | 2-3 hours posttransfusion
  s.Mg
serum iron | 2-3 hours posttransfusion
  s.Fe
serum Calcium | 2-3 hours posttransfusion
  s.Ca

CONTACTS AND LOCATIONS:
Overall Officials: Rania A. El-Farrash, M.D, Study Director — Ain Shams University
Locations (1):
- Rania Farrash, Cairo, Egypt